CLINICAL TRIAL: NCT05403723
Title: A Phase 1b Trial of Adaptive Stereotactic Body Radiotherapy in Combination With Durvalumab (MEDI4736), Platinum, and Etoposide in Extensive Stage Small Cell Lung Cancer
Brief Title: Adaptive SBRT Plus Chemoimmunotherapy for ES-SCLC
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: PI changed institution. Not yet approved at current location.
Sponsor: Taofeek Owonikoko (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Taofeek Owonikoko, Executive Director, University of Maryland Greenebaum Compreshensive Cancer Center, University of Maryland, Baltimore
Organization: University of Maryland, Baltimore (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2464GCCC_HP-00110765
Record Dates: First submitted 2022-05-28; First posted 2022-06-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: Lung Cancer; Chemoimmunotherapy; Stereotactic Body Radiotherapy; Durvalumab; Platinum; Etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — durvalumab; Etoposide; Cisplatin; Platinum; Carboplatin; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Treatment Arm (Experimental): Eligible patients will complete 2 cycles of study treatment with durvalumab, platinum (cisplatin or carboplatin per investigator choice), and etoposide. Patients will then undergo standard of care restaging imaging. Those patients who have a partial or complete response will continue with combination systemic therapy, without additional intervention.
  In patients with less than a partial response (stable disease or progressive disease), SBRT will be given prior to cycle 3 of systemic therapy. The radiotherapy will be given in 5 fractions of 6 Gy to the primary tumor site. See study schema. Patients who undergo SBRT will resume systemic therapy within 2 weeks of completing SBRT and the interval between cycle 2 and cycle 3 should not exceed 6 weeks. Subsequent restaging imaging will continue as per standard of care. All patients will continue maintenance therapy with durvalumab until confirmed progressive disease.
  Interventions: Drug: Durvalumab 50 MG/1 ML Intravenous Solution; Drug: Etoposide Injection; Drug: Cisplatin; Drug: Carboplatin; Device: Stereotactic Body Radiotherapy

INTERVENTIONS:
Drug: Durvalumab 50 MG/1 ML Intravenous Solution — Durvalumab (1500 mg durvalumab via IV infusion) in combination with platinum doublet chemotherapy will be administered to patients once every 3 weeks for up to 4 cycles plus SBRT (platinum resistant group) or without SBRT (platinum sensitive group). Each 3-week of chemoimmunotherapy interval is considered a cycle. Patients with platinum sensitive disease will receive the combination of durvalumab and chemotherapy (total of four cycles) while those with platinum resistant SCLC will receive SBRT and continue to receive up to two additional cycles of treatment with durvalumab along with platinum/etoposide (not to exceed a total of four6 cycles of chemoimmunotherapy including 2 cycles obtained prior to SBRT). Following completion of 4-6 cycles of combination therapy, patients in both groups will continue with maintenance durvalumab (1500 mg) in q4w cycles until disease progression.
Drug: Etoposide Injection — A platinum/etoposide doublet will be administered according to institutional standards. Platinum-etoposide will consist of etoposide 80-100 mg/m2 on days 1-3 of each cycle along with a choice of either carboplatin area under the curve 5-6 mg/mL per min or cisplatin 75-80 mg/m2 (administered on day 1 of each cycle).
Drug: Cisplatin — A platinum/etoposide doublet will be administered according to institutional standards. Platinum-etoposide will consist of etoposide 80-100 mg/m2 on days 1-3 of each cycle along with a choice of either carboplatin area under the curve 5-6 mg/mL per min or cisplatin 75-80 mg/m2 (administered on day 1 of each cycle).
  Other Names: Platinum
Drug: Carboplatin — A platinum/etoposide doublet will be administered according to institutional standards. Platinum-etoposide will consist of etoposide 80-100 mg/m2 on days 1-3 of each cycle along with a choice of either carboplatin area under the curve 5-6 mg/mL per min or cisplatin 75-80 mg/m2 (administered on day 1 of each cycle).
  Other Names: Platinum
Device: Stereotactic Body Radiotherapy — Patients will receive palliative radiation to the primary tumor site up to 30 Gy for 1 week given as 5 daily fractions of 6 Gy each or 27 Gy as 3 fractions of 9 Gy administered every other day.
  Other Names: SBRT

SUMMARY:
This is trial studying the safety of adaptive stereotactic body radiotherapy (SBRT) combined with durvalumab immunotherapy, platinum chemotherapy, and etoposide chemotherapy in platinum refractory extensive stage small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
This is a phase Ib, open-label, single-arm study in newly diagnosed patients with extensive stage SCLC, to test the safety of the adaptive addition of SBRT to combination therapy with durvalumab, platinum, and etoposide. Approximately 50 patients with ES-SCLC will be enrolled in this study in order to identify 20 patients with platinum refractory disease who do not show evidence of early response to chemoimmunotherapy. Eligible patients will complete 2 cycles of study treatment with durvalumab, platinum (cisplatin or carboplatin per investigator choice), and etoposide. Patients will then undergo standard of care restaging imaging. Those patients who have a partial or complete response will continue with combination systemic therapy, without additional intervention.

In patients with less than a partial response (stable disease or progressive disease), SBRT will be given prior to cycle 3 of systemic therapy. The radiotherapy will be given in 5 fractions of 6 Gy to the primary tumor site. See study schema. Patients who undergo SBRT will resume systemic therapy within 2 weeks of completing SBRT and the interval between cycle 2 and cycle 3 should not exceed 6 weeks. Subsequent restaging imaging will continue as per standard of care. All patients will continue maintenance therapy with durvalumab until confirmed progressive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age > 18 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Body weight >30 kg
5. Adequate normal organ and marrow function as defined below:

   1. Hemoglobin ≥10.0 g/dL
   2. Absolute neutrophil count (ANC) ≥1.5 × 109 /L
   3. Platelet count ≥100 × 109/L
   4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
   5. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   6. Creatinine WNL or if >ULN, then measured creatinine clearance (CL) >50 mL/min or calculated creatinine CL>50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
6. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
7. Confirmed histologic or cytologic diagnosis of small cell lung cancer
8. No prior treatment for ES-SCLC (patients who received not more than one cycle of chemotherapy ± durvalumab as SOC prior to enrolment may be allowed on study at the discretion of the study sponsor)
9. Extensive stage disease at diagnosis
10. Measurable disease per Recist 1.1
11. Female Patients must either be of non-reproductive potential (i.e., post-menopausal by history: ≥50 years old and no menses for 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 4 weeks prior to first dose of IP
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any unresolved toxicity National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study PI/Sponsor
4. Major surgical procedure within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
5. History of allogenic organ transplantation.
6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
7. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
8. History of another primary malignancy except for

   1. Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease
9. History of leptomeningeal carcinomatosis
10. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 2-5 minutes apart)
11. History of active primary immunodeficiency
12. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for chemotherapy or hypersensitivity reactions (e.g., CT scan premedication)
14. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
15. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control (see Table 6) from screening to 90 days after the last dose of durvalumab monotherapy.
16. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
17. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
18. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements
19. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) and interstitial lung disease
20. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
21. Symptomatic or uncontrolled brain metastases requiring treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids. (Patients with small untreated but asymptomatic brain lesions are eligible).
22. Patients with uncontrolled seizures.
23. Previous treatment with definitive chemoradiation for LS-SCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (AEs) | Up to 2.5 years
  Number of patients that experience Adverse Events (AEs) assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Adverse Events will be described by Type, Category, including only most severe Grade experienced by a single patient.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2.5 years
  Proportion of patients with objective response (Complete Response (CR) + Partial Response (PR)) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR) is defined as: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is defined as: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, MD, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No